CLINICAL TRIAL: NCT04765345
Title: Rate of Progression of PCDH15-Related Retinal Degeneration in Usher
Brief Title: Rate of Progression of PCDH15-Related Retinal Degeneration in Usher Syndrome 1F
Acronym: RUSH1F
Status: Active, not recruiting | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Usher 1F Collaborative (Unknown); Marjorie C. Adams Foundation (Unknown); Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Other Study IDs: RUSH1F
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Retinal Degeneration; Retinitis Pigmentosa; Eye Diseases, Hereditary
Keywords: PCDH15
MeSH Terms: conditions — Retinal Degeneration; Retinitis Pigmentosa; Eye Diseases, Hereditary; Deafness, Autosomal Recessive 23

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vision Cohort 1: ~25 participants with the better eye Screening Visit visual acuity ETDRS letter score of 54 or more [approximate Snellen equivalent 20/80 or better] and visual field diameter 10 degrees or more in every meridian of the central field.
  The better eye is defined as the eye with better Screening Visit ETDRS VA. If both eyes have the same VA (defined as the same Snellen equivalent), then the determination will be made at investigator discretion as the eye with better fixation or clearer ocular media to permit highest quality retinal imaging.
  The visual field (VF) is defined as the clinically determined kinetic VF III4e performed within the last 18 months prior to or including the Screening Visit date.
- Vision Cohort 2: ~15 participants with the better eye Screening Visit visual acuity ETDRS letter score of 19-53 [approximate Snellen equivalent 20/100 - 20/400] or (visual acuity ETDRS letter score of 54 or more [approximate Snellen equivalent 20/80 or better] and visual field diameter less than 10 degrees in any meridian of the central field).
  The better eye is defined as the eye with better Screening Visit ETDRS VA. If both eyes have the same VA (defined as the same Snellen equivalent), then the determination will be made at investigator discretion as the eye with better fixation or clearer ocular media to permit highest quality retinal imaging.
  The visual field (VF) is defined as the clinically determined kinetic VF III4e performed within the last 18 months prior to or including the Screening Visit date.

SUMMARY:
The overall goal of this project, co-funded by the Foundation Fighting Blindness and the USHER 1F Collaborative is to characterize the natural history of disease progression in patients with PCDH15 mutations in order to accelerate the development of outcome measures for clinical trials.

DETAILED DESCRIPTION:
This natural history study of patients with PCDH15 disease-causing variants will accelerate the development of outcome measures for clinical trials. Sensitive, reliable outcome measures of retinal degeneration will greatly facilitate development of treatments for retinitis pigmentosa due to PCDH15 disease-causing variants. Together these approaches are expected to have an impact on understanding PCDH15 related retinal degeneration, developing experimental treatment protocols, and assessing their effectiveness.

The goals and expected impact of this natural history study are to:

1. Describe the natural history of retinal degeneration in patients with biallelic disease-causing variants in the PCDH15 gene
2. Contribute to the identification of sensitive structural and functional outcome measures to use for future multicenter clinical trials in PCDH15 related retinal degeneration
3. Contribute to the identification of populations for future clinical trials of investigative treatments for PCDH15 related retinal degeneration

Study Objectives

The primary objectives of the natural history study are to:

1. Characterize the natural history of retinal degeneration associated with biallelic pathogenic mutations in the PCDH15gene over 4 years, as measured using functional, structural, and patient-reported outcome measures
2. Explore whether structural outcome measures can be validated as surrogates for functional outcomes in individuals with biallelic pathogenic mutations in the PCDH15 gene
3. Explore possible risk factors (genotype, phenotype, environmental, and comorbidities) for progression of the outcome measures at 4 years in individuals with biallelic pathogenic mutations in the PCDH15 gene
4. Explore variability and symmetry of left and right eye outcomes over 4 years in individuals with biallelic pathogenic mutations in the PCDH15 gene

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following inclusion criteria at the Screening Visit in order to be eligible to enroll into the genetic screening phase.

1. Willing to participate in the study and able to communicate consent during the consent process
2. Ability to return for all study visits over 48 months
3. Age ≥ 8 years
4. Not planning to enroll in an experimental clinical trial for the treatment of PCDH15 for the duration of this study
5. Must meet one of the Genetic Screening Criteria, defined below:

   * Screening Group A: At least 2 disease-causing variants in the PCDH15 gene which are homozygous or heterozygous in trans, based on a report from a clinically certified lab (or a report from a research lab that has been pre- approved by the Genetics Committee)
   * Screening Group B: Only 1 disease-causing variant in the PCDH15 gene, based on a report from a clinically certified lab (or a report from a research lab which has been pre-approved by the Genetics Committee)
   * Screening Group C: At least 2 disease-causing variants in the PCDH15 gene which are unknown phase, based on a report from a clinically certified lab (or a report from a research lab which has been pre-approved by the Genetics Committee)

Note pertaining to all Screening Groups: if a participant has a variant(s) of unknown significance, he/she would still qualify if there is at least 1 disease-causing variant(s) on the PCDH15 gene. The Genetics Committee will review unique cases where segregation analysis is not feasible to determine eligibility.

Ocular Inclusion Criteria

Both eyes must meet all the following at the Screening Visit for a participant to be eligible to enroll into the genetic screening phase.

1. Clinical diagnosis of retinal dystrophy
2. Clear ocular media and adequate pupil dilation to permit good quality photographic imaging

Exclusion Criteria:

Participants must not meet any of the following exclusion criteria at the Screening Visit in order to be eligible to enroll into the genetic screening phase.

1. Mutations in genes that cause autosomal dominant retinitis pigmentosa (ADRP), X-linked retinitis pigmentosa (RP), or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than PCDH15
2. Expected to enter experimental treatment trial at any time during this study
3. History of more than 1 year of cumulative treatment, at any time, with an agent associated with pigmentary retinopathy (including hydroxychloroquine, chloroquine, thioridazine, and deferoxamine)

Note: Pregnant women are not being specifically excluded from participation.

Ocular Exclusion Criteria

If either eye has any of the following at the Screening Visit, the participant is not eligible to enroll into the genetic screening phase.

1. Current vitreous hemorrhage
2. Current or any history of tractional or rhegmatogenous retinal detachment
3. Current or any history of (e.g., prior to cataract or refractive surgery) spherical equivalent of the refractive error worse than -8 Diopters of myopia
4. History of intraocular surgery (e.g., cataract surgery, vitrectomy, penetrating keratoplasty, or LASIK) within the last 3 months
5. Current or any history of confirmed diagnosis of glaucoma (e.g., based on glaucomatous VF changes or nerve changes, or history of glaucoma filtering surgery)
6. Current or any history of retinal vascular occlusion or proliferative diabetic retinopathy
7. History or current evidence of ocular disease that, in the opinion of the investigator, may confound assessment of visual function
8. History or evidence of active treatment for retinitis pigmentosa that could affect the progression of retinal degeneration, including:

   1. Any use of ocular stem cell or gene therapy
   2. Any treatment with ocriplasmin
   3. Treatment with an ophthalmic oligonucleotide within the last 9 months (last treatment date is less than 9 months prior to Screening Visit date)
   4. Treatment with any other product within five times the expected half-life of the product (time from last treatment date to Screening Visit date is at least 5 times the half-life of the given product)
   5. Treatment with Ozurdex (dexamethasone), Iluvien or Yutiq (fluocinolone acetonide) intravitreal implant

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be recruited from approximately 10 clinical sites worldwide. All eligible participants will be included without regard to gender, race, or ethnicity. Potential eligibility will be assessed during a routine examination by an investigator prior to obtaining informed consent, as part of usual care, through referrals from other providers or self-referral.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Field Sensitivity | Baseline (all Vision Cohort 1 and 2 participants will complete two tests at baseline. The results will be compared according to the visual field criteria to determine if a third test is needed), 12Month, 24Month, 36Month, and 48Month
  measured by static perimetry with quantitative, topographic analysis (Hill of Vision) and assessed by a central reading center
Change in Best Corrected Visual Acuity | Screening, Baseline, 12Month, 24Month, 36Month, and 48Month
  Early Treatment of Diabetic Retinopathy Study (ETDRS) Best corrected visual acuity (BCVA) letter score as measured on the Electronic Visual Acuity (EVA) system or ETDRS charts. Letter score range values=0-100 (with higher values = better and lower values = worse.) Berkeley Rudimentary Vision Test (BRVT) will be used for patients unable to see letters.
Change in Mean Retinal Sensitivity | Baseline (all Vision Cohort 1 and 2 participants will complete two tests at baseline. The results will be compared according to the visual field criteria to determine if a third test is needed), 12Month, 24Month, 36Month, and 48Month
  Measured by fundus-guided microperimetry (MP) and assessed by a central reading center at selected sites with requisite equipment.
Change in Full-field Retinal Sensitivity | Baseline, 12Month, 24Month, 36Month, and 48Month
  Measured by full-field stimulus threshold (FST) testing to blue, white and red stimuli.
Change in Best Corrected Low Luminance Visual Acuity (LLVA) | Screening, Baseline, 12Month, 24Month, 36Month, and 48Month
  Measured by Letter Score. Letter score range values=0-100 (with higher values = better and lower values = worse.)
Change in Contrast Sensitivity Function (CSF) | Baseline, 12Month, 24Month, 36Month, and 48Month
  Measured by the CSV-1000E VectorVision chart
Change in ellipsoid zone (EZ) area | Baseline, 12Month, 24Month, 36Month, and 48Month
  Measured by spectral domain optical coherence tomography (SD-OCT) and assessed by a central reading center.

SECONDARY OUTCOMES:
Explore qualitative categorization of Fundus Autofluorescence (FAF) pattern | Baseline, 12Month, 24Month, 36Month, and 48Month
  Assessed by a central reading center.
Explore quantitative measures of FAF | Baseline, 12Month, 24Month, 36Month, and 48Month
  Assessed by a central reading center.

OTHER OUTCOMES:
Patient Reported Outcomes (Adults 18 years or older) | Baseline, 24Month, and 48Month
  Measured by Michigan Retinal Degeneration Questionnaire (MRDQ) MRDQ - consists of 59 items using categories: : ''None: I do not have trouble with this,'' ''A little difficulty: I notice a problem, but I do not struggle,'' ''Moderate difficulty: I struggle but I can still do this,'' ''Extreme difficulty : I struggle a lot and sometimes I cannot do this,'' and ''N/A for non-vision reasons: I do not do this.'
Patient Reported Outcomes (Adults 18 years or older) | Baseline, 24Month, and 48Month
  Measured by Patient-Reported Outcomes Measurement Information System (PROMIS®-29)
Patient Reported Outcomes (less than 18 years): | Baseline, 24Month, and 48Month
  L. V. Prasad-Functional Vision Questionnaire (LVP-FVQ II) The LVP-FVQ II consists of 23 items using 3 categories: 1, no difficulty; 2, some difficulty; 3, a lot of difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Stingl, MD, Study Chair — University Hospital Tuebingen
Locations (10):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - The Johns Hopkins Wilmer Eye Institute, Baltimore, Maryland
  - Duke University, Duke Eye Center, Durham, North Carolina
- Hospital for Sick Children, Toronto, Ontario, Canada
- CHNO des Quinze-Vingts, Paris, France
- University of Tubingen, Tübingen, Germany
- Haddassah Medical Center, Jerusalem, Israel
- Radboud University, Nijmegen, Netherlands
- University Hospital Basel, Basel, Switzerland
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
A de-identified database is placed in the public domain on the FFB/Jaeb public website after the completion of each protocol and publication of the manuscript.
Supporting Information: Study Protocol, ICF
Time Frame: After manuscript is published
Access Criteria: Users accessing data must enter an email address

REFERENCES:
- See also: Foundation Fighting Blindness Public Website — https://public.jaeb.org/ffb

DOCUMENTS (2):
  • Study Protocol: RUSH1F Protocol (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT04765345/Prot_000.pdf
  • Study Protocol: Protocol Administrative Change Letter (PACL) (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT04765345/Prot_001.pdf